CLINICAL TRIAL: NCT04533906
Title: Study to Investigate if Sucking a Coldamaris Lozenge Elutes Sufficient Iota-carrageenan to Inactivate Usual Common Cold Viruses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marinomed Biotech AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LOA_19_04
Record Dates: First submitted 2020-08-21; First posted 2020-09-01 (Actual); Last update posted 2021-01-08 (Actual); Status verified 2020-10

CONDITIONS: Common Cold; Viral Infection
Keywords: respiratory virus; carrageenan; coronavirus; influenza virus; human rhinovirus; coxsackie virus; Carragelose; Iota-carrageenan
MeSH Terms: conditions — Common Cold; Virus Diseases; Coronavirus Infections; Coxsackievirus Infections

STUDY DESIGN:
Intervention Model Description: The saliva of subjects will be collected before and during sucking a Coldamaris lozenge.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Carrageenan (Experimental): Subjects sucking carageenan containing lozenge
  Interventions: Device: Coldamaris lozenges

INTERVENTIONS:
Device: Coldamaris lozenges — sucking carageenan containing lozenge
  Other Names: Betadine; Quixx protect; Quixx grip-protect

SUMMARY:
Coldamaris lozenges are a medical device containing 10 mg carrageenan/lozenge. The goal of the study is to determine whether the iota-carrageenan content in the saliva of subjects who sucked Coldamaris® lozenges is sufficient to inhibit the replication of 4 of the most common respiratory viruses causing common cold. At least 29 subjects will be screened, in order to get 24 subjects included.

DETAILED DESCRIPTION:
Coldamaris lozenges are a medical device containing 10 mg carrageenan/lozenge. The goal of the study is to determine whether the iota-carrageenan content in the saliva of subjects who sucked Coldamaris® lozenges is sufficient to inhibit the replication of 4 of the most common respiratory viruses causing common cold. At least 29 subjects will be screened, in order to get 24 subjects included.

The primary objective is whether the mean iota-carrageenan concentration in saliva during sucking an iota-carrageenan containing lozenge reaches published IC90 values for HRV1a and HRV8.

The secondary objectives are whether the mean iota-carrageenan concentration in saliva (µg/ml; base line corrected) during sucking an iota-carrageenan containing lozenge reaches the respective IC90/MIC values (paired t-tests) of the clinical saliva samples for HRV1a, HRV8, hCoV OC43, influenza virus H1N1n and Coxsackie virus A10.

ELIGIBILITY:
Inclusion Criteria:

* personally signed and dated informed consent
* healthy respiratory tract, no acute infection
* age > 18 years

Exclusion Criteria:

* subjects with signs of an acute respiratory infection
* subjects with a known hypersensitivity to one of the ingredients
* presence of pregnancy confirmed

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2020-08-04 (Actual); Primary Completion 2020-10-04 (Actual); Study Completion 2020-11-10 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure is the iota-carrageenan concentration in saliva. | 3 months
  The mean iota-carrageenan concentration in saliva during sucking an iota-carrageenan containing lozenge should reach published IC90 values for 2 human rhinoviruses.

SECONDARY OUTCOMES:
The secondary outcome measure is the iota-carrageenan concetration in salvia. | 3 months
  Iota-carrageenan concentration in saliva of subjects should be high enough to inhibit replication of human rhinoviruses, human Coronavirus OC43, human influenzavirus H1N1n, and Coxsackievirus A10.

CONTACTS AND LOCATIONS:
Locations (1):
- Dr. Friedrich Ehrenreich, Vienna, Austria

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Morokutti-Kurz M, Unger-Manhart N, Graf P, Rauch P, Kodnar J, Grosse M, Setz C, Savli M, Ehrenreich F, Grassauer A, Prieschl-Grassauer E, Schubert U. The Saliva of Probands Sucking an Iota-Carrageenan Containing Lozenge Inhibits Viral Binding and Replication of the Most Predominant Common Cold Viruses and SARS-CoV-2. Int J Gen Med. 2021 Sep 7;14:5241-5249. doi: 10.2147/IJGM.S325861. eCollection 2021. PMID 34526804